CLINICAL TRIAL: NCT01858233
Title: The IBEP Study: a Randomized Control Trial of an Educational Intervention for Lifestyle Modification in Women With Gestational Diabetes.
Brief Title: The IBEP Study: an Intervention for Lifestyle Modification in Women With Gestational Diabetes
Acronym: IBEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IBEP
Record Dates: First submitted 2013-05-08; First posted 2013-05-21 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Gestational Diabetes; Weight Gain During Pregnancy; Weight Loss After Pregnancy
Keywords: Gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Behavioral Modification (Experimental): intensive dietary counseling, increased activity, lactation consult
  Interventions: Behavioral: Intensive Behavioral Modification
- Routine care (No Intervention): standard dietary counseling

INTERVENTIONS:
Behavioral: Intensive Behavioral Modification — Intensive dietary counseling, increased physical activity, lactation counseling
  Arms: Intensive Behavioral Modification

SUMMARY:
The IBEP study is a randomized control trial of a healthy lifestyle intervention program for women with gestational diabetes. The primary aim of the study is to evaluate whether women with gestational diabetes enrolled in an intensive behavioral educational program (IBEP) demonstrate lower mean fasting glucose levels measured by 2 hour 75 gram oral glucose tolerance test (OGTT) at 6 weeks postpartum compared to women with gestational diabetes who undergo routine gestational diabetes education and counseling.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with gestational diabetes between 20 and 34 weeks gestation

Exclusion Criteria:

* women on chronic steroid therapy
* women with a diagnosis of GDM <20 weeks or >34 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The IBEP Study | 2 years
  To evaluate mean fasting glucose levels measured by 2 hour 75 gram oral glucose tolerance test (OGTT) at 6 weeks in women enrolled in an intensive behavioral educational program compared to women with GDM who undergo routine GDM education and counseling.

SECONDARY OUTCOMES:
The IBEP Study | 2 years
  To evaluate the amount of weight lost in women enrolled in an intensive behavioral program and whether it correlates with more favorable lipid profiles at 6 weeks postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Durnwald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Durnwald CP, Kallan MJ, Allison KC, Sammel MD, Wisch S, Elovitz M, Parry S. A Randomized Clinical Trial of an Intensive Behavior Education Program in Gestational Diabetes Mellitus Women Designed to Improve Glucose Levels on the 2-Hour Oral Glucose Tolerance Test. Am J Perinatol. 2016 Oct;33(12):1145-51. doi: 10.1055/s-0036-1585085. Epub 2016 Jul 11. PMID 27398697